CLINICAL TRIAL: NCT07048925
Title: Endovascular Treatment of TASC II C-D Iliac Artery Lesions Using Covered Stents: A Retrospective Cohort Study
Brief Title: Iliac Stent-Grafts in TASC C-D Lesions
Status: Active, not recruiting | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: SUKAEK-2023/01/08
Record Dates: First submitted 2025-06-14; First posted 2025-07-03 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-06

CONDITIONS: Aortoiliac Occlusive Disease; Endovascular Treatments; Peripheral Arterial Disease(PAD)
Keywords: TASC C-D Lesions; Iliac Stent-Graft; Non-Surgical Revascularization; Covered Stents
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the midterm outcomes of patients with advanced aortoiliac artery narrowing (TASC C-D lesions) who were treated with covered iliac stent-grafts instead of open surgery. These patients were either too high-risk for surgery or refused it. Medical records from the past five years at a single cardiovascular surgery center in Turkey were reviewed retrospectively. The research focuses on the success rate of the procedure, complications, vessel patency, and the need for additional treatments. The results may help guide treatment decisions in similar high-risk patients who are not candidates for open vascular surgery.

DETAILED DESCRIPTION:
This is a single-center retrospective cohort study evaluating intermediate-term outcomes of patients with aortoiliac occlusive disease who underwent endovascular treatment using covered iliac stent-grafts. The study includes patients with complex iliac artery lesions (typically classified as TASC II C or D) treated over the past five years. Open surgery was not feasible or preferred in these cases due to high surgical risk or patient refusal.The study analyzes medical records to assess technical success, symptom improvement, complication rates, vessel patency, and the need for reintervention. Results may inform the role of covered stent-grafts as a viable alternative in managing advanced aortoiliac disease in high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with TASC C-D iliac artery lesions
2. Procedures done within last 5 years in the same clinic
3. Aged between 18-85 years
4. Not eligible for open surgery or refused it

Exclusion Criteria:

1. TASC A-B lesions
2. Age <18 or >85

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with peripheral artery disease and TASC C-D iliac lesions treated with covered stents between 2018 and 2023
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Technical and Clinical Success of Covered Iliac Stent-Graft | Within 5 years before the study start
  Based on review of patient records over the past 5 years, including procedural success and symptom relief

SECONDARY OUTCOMES:
Complications, Patency Rates, and Reintervention Needs | Within 5 years before the study start
  Post-procedural outcomes such as restenosis, thrombosis, or need for surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Emrah Ereren, Study Chair — Samsun University Faculty of medicine
Locations (1):
- Samsun University Faculty of Medicine, Samsun, Turkey (Türkiye)